CLINICAL TRIAL: NCT06024967
Title: The Safety and Efficacy of Once-weekly PEG-somatropin (GenSci004) in Children With Growth Hormone Deficiency: An Open-label, Single-arm, Multicenter Phase 3 Study
Brief Title: A Study to Investigate the Safety and Efficacy of Once-weekly PEG-somatropin (GenSci004) in Children With Growth Hormone Deficiency
Acronym: ESCALATE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci004-302
Record Dates: First submitted 2023-08-09; First posted 2023-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: GHD
Keywords: GHD; growth hormone deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- GenSci004 (Experimental)
  Interventions: Drug: PEG-somatropin

INTERVENTIONS:
Drug: PEG-somatropin — PEG-somatropin

SUMMARY:
The purpose of this Phase 3 study is to evaluate the safety and efficacy of once-weekly GenSci004 over 108 weeks in children with GHD aged from 6 months to 17 years old, inclusive.

DETAILED DESCRIPTION:
The purpose of this Phase 3 study is to evaluate the safety and efficacy of once-weekly GenSci004 over 108 weeks in children with GHD aged from 6 months to 17 years old, inclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Investigator-determined diagnosis of GHD prior to the historical initiation of daily rhGH trerapy
2. Participant must be 6 months to 17 years old
3. Tanner stage <5 at Visit 1
4. Open epiphyses
5. Normal fundoscopy at Screening
6. Written, signed, informed consent of the participant's parent(s)/LAR(s) and written assent of the participant

Exclusion Criteria:

1. History or presence of malignant disease
2. Children with diabetes mellitus
3. Major medical conditions and/or presence of contraindications to GH treatment
4. Pregnancy
5. Participation in any other study of an investigational agent within three months prior to Visit 1
6. Prior exposure to investigational drug or any other long-acting growth hormone
7. Any other reason per investigator's discretion

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events of once-weekly GenSci004 in children with GHD | 108 weeks
  Incidents of adverse events

SECONDARY OUTCOMES:
Annualized Height Velocity (AHV) | 104 weeks
  Measured in centimeter per year (cm/year)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Silverman, MD, Study Chair — Morristown Medical Center

IPD SHARING:
Plan to Share IPD: Yes